CLINICAL TRIAL: NCT04608981
Title: Effect of Diclofenac Potassium Versus Prednisolone as a Premedication on Post-endodontic Pain and Pulpal Interleukin (IL)-8 Expression in Symptomatic Irreversible Pulpitis Cases: A Randomized Clinical Trial
Brief Title: Effect of Diclofenac Potassium Versus Prednisolone on Post-endodontic Pain and Pulpal IL-8 Expression
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Adel Abdullah Ali Soliman, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CairoU_IL8
Record Dates: First submitted 2020-10-13; First posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Symptomatic Irreversible Pulpitis
Keywords: prednisolone; diclofenac potassium; interleukin-8
MeSH Terms: interventions — Prednisolone; Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In this proposed study, the participant, and the assessor will be blinded. The participants will be blinded to the study hypothesis as to which intervention is expected to be better.
  The patients, who already do not know their treatment group, will assess the level of their post-endodontic pain.
  * The laboratory technician at the microbiological department will not know the treatment group of the patients.
  * The treatment groups will remain anonymous at the end of the study during assessment by the statistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Prednisolone premedication (Experimental): Single, oral dose of 30 mg prednisolone pre-medication 30 min before starting endodontic treatment.
  Interventions: Drug: Prednisolone 30 mg
- Diclofenac potassium premedication (Experimental): Single, oral dose of 50 mg diclofenac potassium pre-medication 1 hour before starting endodontic treatment.
  Interventions: Drug: Diclofenac Potassium 50mg Tab
- Placebo (Placebo Comparator): Placebo tablet 1 hour before starting endodontic treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prednisolone 30 mg — Steroidal anti-inflammatory drug as a preoperative medication
  Other Names: One and a half tablets Solupred oro 20 mg, ARE, Aventis Intercontinental, Paris, France
  Arms: Prednisolone premedication
Drug: Diclofenac Potassium 50mg Tab — Non-steroidal anti-inflammatory drug as a preoperative medication
  Other Names: Cataflam; NOVARTIS Pharma, Basel, Switzerland
  Arms: Diclofenac potassium premedication
Drug: Placebo — Starch
  Arms: Placebo

SUMMARY:
To assess the effect of using diclofenac potassium versus prednisolone as a pre-medication compared to placebo on:

* Intensity of post-endodontic pain in patients with symptomatic irreversible pulpitis.
* Pulpal IL-8 expression.
* Incidence of post-endodontic pain in patients with symptomatic irreversible pulpitis.

DETAILED DESCRIPTION:
After confirming the diagnosis and making sure that the patient conforms to all eligibility criteria, the principal investigator will enroll the patient in the study.

* Patients will be asked to rate their pre-operative pain intensity (ie, before the commencement of any treatment [baseline score]; on the visual analogue scale "VAS"
* Enrolled patients will be randomly assigned into one of three groups:

Intervention Group 1 (Diclofenac Potassium): single, oral dose of 50 mg diclofenac potassium pre-medication (Cataflam; NOVARTIS Pharma, Basel, Switzerland) one hour before starting endodontic treatment.

Intervention Group 2 (Prednisolone): single, oral dose of 30 mg prednisolone (one and a half tablets Solupred oro 20 mg, ARE, Aventis Intercontinental, Paris, France) 30 min before starting endodontic treatment.

Control Group (Placebo): The patients assigned to this group will be given a placebo tablet (Starch, Bridgewater, NJ) one hour before starting endodontic treatment.

- Root canal therapy in all groups will be completed by the principal investigator in a single visit as follows:

1. Anesthetizing the tooth using inferior alveolar nerve block technique by local anesthesia of 1.8 ml of 2% Mepivacaine HCl with 1:100,000 epinephrine.
2. After anesthesia is achieved and verified with Endo-Ice, the patient's tooth is isolated with a rubber dam, caries is excavated, and the pulp is exposed with a sterile round bur.
3. Preparation of access cavity using a sterile round carbide bur and an Endo-Z bur
4. Sample Collection:

   * Blood from the exposed surface of the pulp will be collected with 2 sterile cotton pellets.
   * The pellets will be held at the exposure site for 45-60 seconds to allow absorption of the blood from the pulpal tissue.
   * The pellets will be placed in 1.0 mL saline in heparin-coated tubes.
   * Samples will be placed on ice and stored/refrigerated immediately at -20 degrees celsius until they are ready to be tested.
5. After the pulpal blood sample is collected, patency of the root canals will be confirmed using stainless steel hand K-files sizes #10 and #15.
6. Working length will be determined using an electronic apex locator then confirmed radiographically to be 1 mm shorter than radiographic apex.
7. Mechanical preparation will be completed in a crown down technique with ProTaper Next10 rotary files set on an endodontic motor adjusted at a speed of 300 rpm and torque of 200 gcm. In-and-out motions will be applied with stroke lengths not exceeding 3mm in the cervical, middle, and apical thirds until attaining the established WL.
8. The root canal will be thoroughly irrigated with 3 mL of 2.6% sodium hypochlorite using a plastic disposable syringe with a 30-gauge side-vented needle reaching 1mm short of the working length between every subsequent instrument, whereas saline will be used as the final irrigant.
9. The canal will then be dried using sterile paper points. Master cone fit radiograph will be taken and then the root canal will be obturated at the same appointment with matching-size gutta percha points and resin-based sealer using cold lateral compaction technique.
10. Access cavity will be sealed with Coltosol F temporary filling material.
11. At the end of the session, each patient will be instructed to complete a pain diary, (VAS), at specific intervals; immediately after treatment completion; and 6, 12, 24, and 48 hours after the completion of treatment. The patient will be asked to mark the level of pain on this 10-cm line. The distance from the left end to the mark made by the patient, which will be measured by the operator with a ruler, is the pain intensity.
12. Patients will be contacted by their operator at each time-point to check on them and as a reminder. Then, information will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-50 years.
* Males and females.
* American Society of Anesthesiologists class 1 or 2.
* Mandibular premolar teeth with:

  * Endodontic pulpal diagnosis of symptomatic irreversible pulpitis
  * Normal/slight widening in the periodontal membrane space (PMS).
* Patients who had not taken any anti-inflammatory drugs the day of the root canal procedure unless they belong to one of the intervention groups.
* Patients who accept to participate in the trial, understand the VAS, and can sign the informed consent

Exclusion Criteria:

* Cases with acute peri-apical conditions (acute apical periodontitis/ acute apical abscess), pulpal necrosis, previously initiated therapy, or previously treated.
* Teeth other than single-rooted teeth.
* Radiographic evidence of external or internal root resorption vertical root fracture, perforation, or calcification.
* Immature teeth.
* Unrestorable teeth or teeth with severe periodontal disease.
* Patients with a known allergy, sensitivity, or history of other adverse reactions to the medications administered.
* Patients with a history of active peptic ulcer within the preceding 12 months, bleeding problems, anticoagulant use within the last month, or kidney disease.
* Patients who took analgesics/ anti-inflammatory drugs (steroidal or non-steroidal) the day of endodontic treatment.
* Pregnant or nursing females.
* Patients who are unable to provide informed consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Change in the intensity of post-endodontic pain | Immediately after treatment completion; and at 6, 12, 24, and 48 hours post-operatively
  Pain intensity will be evaluated using visual analogue scale

SECONDARY OUTCOMES:
Quantification of pulpal IL-8 | During the procedure
  Il-8 analasys will be done via enzyme-linked immunosorbent assay (ELISA)

OTHER OUTCOMES:
Change in the incidence of post-endodontic pain | Immediately after treatment completion; and at 6, 12, 24, and 48 hours post-operatively
  Pain incidence will be evaluated using visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Soliman, MSc, Principal Investigator — Cairo University; Khaled Ezzat, PhD, Study Director — Cairo University; Sara S Abouelenien, PhD, Study Chair — Cairo University

IPD SHARING:
Plan to Share IPD: No